CLINICAL TRIAL: NCT02150902
Title: AUGMENTED WIDE AREA CIRCUMFERENTIAL CATHETER ABLATION FOR REDUCTION OF ATRIAL FIBRILLATION RECURRENCE - A RANDOMIZED CLINICAL TRIAL (The AWARE Trial)
Brief Title: Augmented Wide Area Circumferential Catheter Ablation for Reduction of Atrial Fibrillation Recurrence
Acronym: AWARE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRIS 2771; 201610PJT-376677 (Other Grant/Funding Number: CIHR)
Record Dates: First submitted 2014-05-27; First posted 2014-05-30 (Estimated); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Atrial Fibrillation
Keywords: Catheter ablation for atrial fibrillation; treatment for atrial fibrillation; comparison of catheter ablation techniques for atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Augmented- WACA (Experimental): Augmented- wide area circumferential catheter ablation for atrial fibrillation
  Interventions: Procedure: Augmented- wide area circumferential ablation procedure
- WACA (Active Comparator): Wide area circumferential catheter ablation procedure for atrial fibrillation
  Interventions: Procedure: Wide area circumferential catheter ablation

INTERVENTIONS:
Procedure: Wide area circumferential catheter ablation — All subjects in the control arm of the trial will undergo wide area circumferential catheter ablation (WACA; lesions delivered 1-2 cm away from the pulmonary vein ostium) around all four pulmonary veins to the endpoint of electrical isolation (demonstrated by entry and exit block using differential pacing). Catheter ablation will be performed using contact force (CF) and electroanatomical mapping system guidance (average CF >10g, FTI > 500 g-sec and minimum ablation duration >10 sec). Dormant pulmonary vein conduction will be tested using adenosine, after completion of the lesion set, and additional lesions will be delivered to eliminate dormant PV conduction.
  Other Names: WACA
  Arms: WACA
Procedure: Augmented- wide area circumferential ablation procedure — Subjects in this group will have WACA performed as described for WACA. Following completion of the WACA procedure a second set of circumferential ablation lesions will be delivered around the first set of ablation lesions. The ablation catheter tip will be positioned at each of the ablation lesions along the first WACA line and then moved away (from the PV ostia) until healthy, non ablated tissue is recorded from the catheter tip. Energy will be delivered using CF and FTI data as described previously. Once the first WACA ablation line has been completely duplicated the procedure will be deemed complete. In case PV isolation is not achieved after the first WACA lesion set repeat electrophysiologic testing will be performed to determine whether the augmented-WACA procedure was successful in achieving PV isolation.
  Other Names: Augmented WACA
  Arms: Augmented- WACA

SUMMARY:
Atrial fibrillation (AF) is an abnormal heart rhythm in which the top chambers of the heart beat very fast. AF catheter ablation is a known technique to convert heart rhythm from AF to normal rhythm. The technique sends out electrical energy through a catheter (long thin round solid tubes) to destroy the heart tissues in a focused area where AF is starting. This technique is practiced at many hospitals, including the Heart Institute, and is not experimental.

The AWARE study will compare two techniques of AF catheter ablation:

1. Ablation of tissues in wide circular bands around the opening of the pulmonary veins (bring blood back from lungs) in the left upper chamber of the heart. A medicine called adenosine will be given to unmask any incompletely ablated area. Additional ablations will be given if required. This is standard procedure.
2. Same as above but adenosine will not be used. Instead, additional ablation of a second circular band of tissues around the opening of the pulmonary veins will be given. This additional ablation is not standard procedure and is considered experimental.

The Investigators are testing if adding more ablation sites will help maintain normal heart rhythm and reduce the rate of return to AF. The study will compare the occurrence of medical events and complications between the two groups.

Identical supplies and equipment used in both techniques have been approved by Health Canada. Adenosine is currently approved by Health Canada for the treatment and diagnosis of arrhythmias.

396 participants from study sites across Canada will be randomly assigned "similar to flipping a coin" to treatment group 1 or group 2.

After the ablation, participants will have study follow-up at 3, 6 and 12 months. All participant's will be followed for a minimum of 12 months.

DETAILED DESCRIPTION:
Clinical relevance:

The problem of PV reconnection and recurrent AF after catheter ablation for paroxysmal AF is one of the important challenges faced by treating physicians.

Rationale:

The understanding of the role contact force plays in adequate lesion formation during catheter ablation and the fact that this may reduce pulmonary vein (PV) reconnection and AF recurrence is an exciting advance in the field of catheter ablation for AF. A few small clinical trials have demonstrated the safety and feasibility of contact force guided catheter ablation in reducing PV reconnection and AF recurrence. There is a clear need for well designed and adequately powered clinical trials to evaluate the effectiveness of this new strategy. The investigators have developed a novel "augmented" CF guided augmented ablation strategy and will test this against the current clinical gold standard ablation technique.

Objective:

Using contact force (CF) technology, our intention is to evaluate an "augmented- wide area circumferential catheter ablation strategy" that could potentially reduce the incidence of pulmonary vein reconnection and AF recurrence after catheter ablation in patients with paroxysmal AF.

Hypothesis:

In patients with symptomatic paroxysmal AF an augmented-wide area circumferential catheter ablation strategy will result in fewer electrocardiographically documented atrial arrhythmias (AF, atrial flutter and atrial tachycardia) recurrences compared to conventional wide-area catheter ablation.

All subjects in the control arm of the trial will undergo wide area circumferential catheter ablation (WACA; lesions delivered 1-2 cm away from the pulmonary vein ostium) around all four pulmonary veins to the endpoint of electrical isolation (demonstrated by entry and exit block using differential pacing). Catheter ablation will be performed using CF and VISITAG guidance (average CF >10g, Force time integral (FTI) > 500 g-sec and minimum ablation duration >10 sec). Dormant PV conduction will be tested using adenosine, after completion of the lesion set, and additional lesions will be delivered to eliminate dormant PV conduction.

In the experimental arm of the trial all subjects will undergo WACA as described above; however without adenosine testing. In addition these subjects will receive "augmented" ablation lesions, guided by CF feedback, on the outer aspect of the first WACA lesion set. Our hypothesis is that this "belts and suspender" strategy of redundant, CF guided antral ablation lesions will result in a wider band of irreversible atrial muscle and cardiac autonomic ganglionated-plexi damage. It is our expectation that the augmented WACA strategy will result in more durable PV isolation and thereby significantly reduce AF recurrence.

Trial Design:

This trial is a multicentre, prospective, randomized, blinded endpoint trial (PROBE) design. Subjects who satisfy the inclusion and exclusion criteria will be enrolled in the clinical trial. Subjects will be randomized (1:1) to either the control arm (WACA only) or the experimental arm (augmented- WACA). Patients randomized to the experimental arm will go on to have augmented-WACA. The first 90 days after catheter ablation will be considered a "blanking-period" and atrial tachyarrhythmias (AF, Atrial Flutter [AFl] or Atrial Tachycardia [AT]) occurring during this period will be documented. However, these will not be considered treatment failures. Patient accrual will occur over a 24-month period and each subject will have a minimum follow-up period of 12 months. The total duration of the trial will be 36-months (24 months for accrual and a minimum of 12 months of follow up for each subject). Patients will be followed at 3, 6, and 12 months, with 14 day continuous ambulatory ECG monitoring done at each follow up visit. A total of three questionnaires will be administered throughout the study, each at a specific time point. The Quality of Life (EQ-5D) and CCS-Severity of AF scale will be completed together, prior to ablation and at the final follow-up visit. The patient satisfaction score will be completed at the final follow-up visit. All participants will be followed for a minimum of 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Subjects must have symptomatic Paroxysmal AF that is refractory to at least one class I or Class III antiarrhythmic medication OR be intolerant of antiarrhythmic medications OR prefer not to trial antiarrhythmic medications
3. At least one episode of AF documented on 12-lead ECG, Holter monitor or Loop recorder.
4. Subjects must be able to provide informed consent

Exclusion Criteria:

1. Subjects with persistent or permanent AF
2. History of previous catheter or surgical ablation for AF
3. Presence of known intracardiac thrombus
4. Subjects with contraindication to systemic oral anticoagulation therapy, including a history of Heparin Induced Thrombocytopenia
5. Subjects with reversible causes of AF
6. Subjects with significant valve disease (moderate or severe mitral/aortic stenosis or regurgitation)
7. Subjects with known adverse reaction to adenosine
8. Subjects with congenital heart disease
9. Subjects that are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 411 (Actual)
Dates: Start 2015-03; Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Time to First Recurrence of any ECG documented AF, AFl or AT | between days 91 and 364 after catheter ablation
  Time to first recurrence of any ECG documented AF, AFl or AT (symptomatic or asymptomatic) occurring between days 91 and 364 after catheter ablation in the absence of Class I or III antiarrhythmic drug therapy.

SECONDARY OUTCOMES:
The need for repeat catheter ablation procedure | days 91 and 364 after catheter ablation
  The need for repeat catheter ablation procedure because of documented recurrence of symptomatic AF, AFl or AT
ECG documented AF | during the first 90 days after catheter ablation
  Incidence of any ECG documented AF (symptomatic or asymptomatic) during the first 90 days after catheter ablation
emergency department visits or hospitalizations | from randomization to day 364
  The need for emergency department visits or hospitalizations
procedure related complications | from ablation to day 364
  Composite safety endpoints- procedure related complications (Stroke, PV stenosis, Pericarditis, Cardiac perforation, Atrio-esophageal fistula, Major bleeding) and/or death.
Quality of Life measurement using (EQ-5 and Canadian Cardiovascular Society-Severity of AF scales) | from randomization to day 364
  Quality of Life (EQ-5 and Canadian Cardiovascular Society-Severity of AF scales)
Total procedure duration | day of the ablation procedure
  total ablation procedure duration in minutes
Total radiation exposure during the procedure | day of the ablation procedure
  Dose area product in McGy.cm2 and cumulative skin dose in mGv
Health Economic Analysis | from randomization to day 364
  Health care related costs

CONTACTS AND LOCATIONS:
Overall Officials: Girish Nair, MD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (11):
- Canada (11):
  - University of Calgary-Foothills Campus, Calgary, Alberta
  - Victoria Cardiac Arrhythmia Trials Inc., Victoria, British Columbia
  - QE II Health Sciences Centre, Halifax, Nova Scotia
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - St. Michael"s Hospital, Toronto, Ontario
  - Toronto General Hospital-University Health Network, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - McGill University Health Center, Montreal, Quebec
  - CIUSSSNIM-Hopital du Sacre-Coeur de Montreal, Montreal, Quebec
  - Institut universitaire de cardiologie et de pneumologie de Quebec, Québec, Quebec
  - Centre hospitalier universitaire de Sherbrooke (CHUS), Sherbrooke, Quebec

REFERENCES:
- [Derived] Nair GM, Birnie DH, Nery PB, Redpath CJ, Sarrazin JF, Roux JF, Parkash R, Bernier M, Sterns LD, Sapp J, Novak P, Veenhuyzen G, Morillo CA, Singh SM, Sadek MM, Golian M, Klein A, Sturmer M, Chauhan VS, Angaran P, Green MS, Bernick J, Wells GA, Essebag V. Standard vs Augmented Ablation of Paroxysmal Atrial Fibrillation for Reduction of Atrial Fibrillation Recurrence: The AWARE Randomized Clinical Trial. JAMA Cardiol. 2023 May 1;8(5):475-483. doi: 10.1001/jamacardio.2023.0212. PMID 36947030
- [Derived] Nair GM, Birnie DH, Wells GA, Nery PB, Redpath CJ, Sarrazin JF, Roux JF, Parkash R, Bernier M, Sterns LD, Novak P, Veenhuyzen G, Morillo CA, Singh SM, Sturmer M, Chauhan VS, Angaran P, Essebag V. Augmented wide area circumferential catheter ablation for reduction of atrial fibrillation recurrence (AWARE) trial: Design and rationale. Am Heart J. 2022 Jun;248:1-12. doi: 10.1016/j.ahj.2022.02.009. Epub 2022 Feb 24. PMID 35219715